CLINICAL TRIAL: NCT00149721
Title: Anterior Pituitary Function in Patients With Hydrocephalus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eli Lilly and Company (Industry)
Organization: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B9R-US-X041 (terminated)
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: hydrocephalus; pituitary function; shunting
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus

INTERVENTIONS:
Procedure: Ventriculo-peritonal shunting

SUMMARY:
Hydrocephalus (secondary or idiopathic) is a condition characterized by dilatation of the lateral and third ventricles, and often associated with increased intracranial pressure (ICP). We hypothesize that either the ventricle dilatation or the increased ICP may cause disturbances in the hypothalamic-pituitary axis, resulting in different degrees of hypopituitarism. The goal of this study is to determine the prevalence of hypopituitarism in adult patients with hydrocephalus.

DETAILED DESCRIPTION:
The Johns Hopkins Adult Hydrocephalus Program evaluates approximately 250 new patients per year for hydrocephalus and associated disorders, resulting in the new diagnosis of hydrocephalus in about 100 patients annually. After treatment with either shunt surgery or third ventriculostomy, virtually all patients are followed on a regular basis by physicians in the program (Dr. Michael Williams, neurologist, and Dr. Daniele Rigamonti, neurosurgeon, both involved in this project).

These patients represent an ideal cohort to study the effect of hydrocephalus on anterior pituitary function. In addition, as data on intracranial pressure is available for all of them, evaluation of pituitary function would allow us to determine whether the level of intracranial pressure correlates with the likelihood of pituitary failure.

We propose to study 20 subjects of both sexes with NPH, aged 18-80 years over a period of 18 months. They will be recruited by direct advertising among the patients cared for by the Adult Hydrocephalus Program. Patients with hydrocephalus will be studied twice (6-12 months apart) whether or not they undergo shunting.

STUDY PROTOCOL:

1. In addition to the comprehensive neurological history and physical examination, further history will be obtained, with particular attention to sexual function and libido in males and menstrual history in women of fertile age, will be collected.
2. After overnight fasting, an indwelling catheter will be inserted in a peripheral vein. Blood for baseline hormonal evaluation (8-9 AM) including: serum free T4 (FT4), TSH, cortisol, GH, IGF-1, prolactin, LH, FSH, Estradiol (in females) and total testosterone (in males). Menstruating females will be studied during follicular phase. Serum IGF-1, testosterone, estradiol and gonadotropin levels will be interpreted in accordance with the patients' age.
3. All subjects will undergo GH stimulation test by combination of GHRH (1 mcg/kg bolus) and arginine (0.5 gm/kg over 30', maximal dose 30 gm). Blood will be dawn at time 30', 60', 90' and 120' after the GHRH bolus injection. The GHRH+arginine test is the most widely used test to determine GH reserve in adults, independently from their age (14). Normal response is a peak serum GH > 9 ng/ml. Both GHRH and arginine are FDA-approved for this purpose, and have no significant side effects (GHRH may cause transient itching and flushing).
4. An AM cortisol below 5 mcg/dl will be considered diagnostic of adrenal insufficiency. Conversely, a value above 15 mcg/dl will be interpreted as indicating normal adrenal function. For serum cortisol values between 5 and 15 mcg/dl, subjects will be studied on a separate day by low-dose (1 mcg) ACTH stimulation test. Blood for serum cortisol measurement will be obtained at baseline and after 30' from ACTH injection. The low-dose ACTH stimulation test is safe, easy to perform, has high sensitivity for partial secondary adrenal insufficiency, and has been recently used in patient with TBI. Normal response is a serum cortisol at 30' > 18.0 mcg/dl.

Subjects who have shunt surgery will undergo a second study of pituitary function not earlier than 6 months and no later than 1 year from the procedure. We will identify the degree of clinical improvement by documenting change in gait with the Tinetti Gait Assessment Tool, and change in dementia with the Mini-Mental-Status exam. If there is sufficient sample size in the clinically improved and unimproved patients, we will compare between-group results.

Patients who have been on systemic glucocorticoids (GC) for longer than 3 weeks during the previous 12 months will be excluded, as GC may cause suppression of hypothalamic-adrenal axis. In subjects who are on phenytoin, unbound T4 will be measured by equilibrium dialysis, as phenytoin may interfere with direct unbound T4 measurement. Subjects already on L-thyroxine replacement will be excluded.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of idiopathic hydrocephalus, made by clinical and CT or MRI imaging demonstrating ventricular dilation, and confirmed by an established protocol of continuous CSF drainage via spinal catheter. Patients who are found to be eligible for VP shunt insertion on the basis of improvement in cognition/psychomotor speed, gait, or urinary continence are referred for surgery

Exclusion Criteria:

Known peripheral gland failure (primary hypogonadism, primary adrenal insufficiency, primary hypothyroidism); known history of pituitary tumor, pituitary surgery, pituitary hemorrhage, brain irradiation, or of identified causes of secondary hydrocephalus (subarachnoidal bleeding, meningitis, encephalitis, head trauma).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2007-12

PRIMARY OUTCOMES:
anterior pituitary function

SECONDARY OUTCOMES:
well being

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Salvatori, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- GCRC Johns Hopkins University, Baltimore, Maryland, United States